CLINICAL TRIAL: NCT07045974
Title: Effects of Mulligan Mobilization and Stretching on Cervical Radiculopathy
Brief Title: Mulligan Mobilization & Stretching Effects of Cervical
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC-01012 Mahnoor Ali
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cervical Radiculopathy
Keywords: Pain; Disability Level; Range of Motion
MeSH Terms: conditions — Radiculopathy; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Mulligan Mobilization (Experimental): Mulligan SNAGs mobilization technique was applied at level C4/5.
  Interventions: Other: Group A-Mulligan Mobilization
- Group B-Stretching Exercises (Experimental): Cervical stretching exercises will be performed.
  Interventions: Other: Group B-Stretching Exercises

INTERVENTIONS:
Other: Group A-Mulligan Mobilization — Group A will receive Mulligan mobilizations (SNAGs). Mulligan SNAGs mobilization technique was applied at level C4/5. Subjects were placed in sitting position and therapist stood behind the patient with therapist's thumbs on spinous process of particular vertebra. Mobilization was given by active movement followed by passive overpressure based on the movement restricted. The duration of treatment was three sets of ten repetitions each.
  Conventional treatment include the following:
  Subjects in both the groups were treated with hot pack (20 min), TENS (2 to 10 Hz), and manual traction along with deep neck flexor, and isometric neck strengthening.
  Arms: Group A-Mulligan Mobilization
Other: Group B-Stretching Exercises — Group B will receive stretching exercises. Subject was asked to lie supine on the plinth and the head was held at the edge of the plinth by the therapist. Then with one hand the therapist held the neck in cervical lateral flexion to the opposite side so as to achieve the stretching of the trapezius muscle. Myofascial release by applying sustained finger pressure for 5-10 s on the involved trapezius was given. A gentle myofascial stretching force was applied to take up slack and sustained until a release occurred. This protocol comprised four sets of 15 stretches with 3 min rest.
  Conventional treatment include the following:
  Subjects in both the groups were treated with hot pack (20 min), TENS (2 to 10 Hz), manual traction along with deep neck flexor, and isometric neck strengthening.
  Arms: Group B-Stretching Exercises

SUMMARY:
1. To evaluate the effectiveness of mulligan mobilization and stretching exercises in reducing pain in individuals with cervical radiculopathy.
2. To evaluate the effectiveness of mulligan mobilization and stretching exercises in reducing disability in individuals with cervical radiculopathy.
3. To evaluate the effectiveness of mulligan mobilization and stretching exercises at improving ranges in individuals with cervical radiculopathy.

DETAILED DESCRIPTION:
Cervical Radiculopathy is a condition characterized by dysfunction of cervical spinal nerve roots which occurs as a result of compression or inflammatory pathology from a space occupying lesion such as a disc herniation, decreased disc height and degenerative changes of the uncovertebral joints anteriorly and zygoapophyseal joints posteriorly. Cervical radiculopathy constitutes 5%-36% of all radiculopathies. In general, rate of occurrence of cervical radiculopathy is 83/100,000 with an increased prevalence in the fifth decade of life (203/100,000).

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  * Both genders
  * Age between 20-50 years
  * Subjects with neck pain radiating down to the arm
  * Patients with positive findings for spurling test, Upper Limb Tension Test (ULTT), cervical distraction test and cervical rotation test towards the symptomatic side
  * Subjects who were willing to participate in the study and willing to take treatment for cervical radiculopathy.

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.

  * Systemic disease potentially affecting the musculoskeletal system Patients experiencing primary shoulder or upper extremity problem of local origin
  * Patients with any cardiovascular disorders and respiratory disorders
  * Patients with any other pathological conditions involving cervical spine like vertebro basilar insufficiency and canal stenosis
  * Patients having osteophytes in cervical vertebrae
  * Patients who were undergoing treatment for neck pain with other means of physiotherapy at the time of the study
  * Hypermobile joints of cervical vertebrae, Cervical fractures, spinal surgery or other spinal pathologies (i.e. ankylosing spondylitis, spondylolysthesis)
  * Peripheral nerve lesions like neurotemesis and axonotemesis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Cervical Pain Intensity Measured by Numeric Pain Rating Scale (NPRS) | 4 Weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable") High test-retest reliability has been observed in both literate and illiterate patients with rheumatoid arthritis (r = 0.96 and 0.95, respectively) before and after medical consultation.
Cervical Range of Motion by Inclinometer | 4 Weeks
  An inclinometer is a device used to measure angles. It is commonly used in physiotherapy to measure the range of motion (ROM) of joints and very similar to a goniometer.
  The digital inclinometer demonstrated excellent reliability (ICC=0.75-0.86), except for the right lateral flexion (ICC=0.74) and left rotation (ICC=0.72).
Cervical Disability by Neck Disability Index (NDI) | 4 Weeks
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.
  Score: /50 Transform to percentage score x 100 = %points. It has 7 items for daily living, 2 for pain and 1 for concentration. Each item is rated from 0 to 5. Total score is presented in percentage. Higher score tells greater disability while 0 means no disability(16).Total score is 50. In cervical radiculopathy patients it has moderate test retest reliability ICC= 0.68 (22).The NDI has a fair to moderate test-retest reliability in patients with mechanical neck pain but also for patients with cervical radiculopathy. The NDI has a good construct validity.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Sadiq, MSPT (OMPT), Principal Investigator — Riphah International University
Locations (1):
- Leady Reading Hospital (LRH), Hayatabad Medical Complex (HMC), Peshawar, KPK, Pakistan